CLINICAL TRIAL: NCT04262310
Title: Standardizing Method and Development of Normal Values to Measure Human Small Intestinal and Colonic Permeability
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 19-008541
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples for permeability measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Aims: To obtain normative data (median, 10th and 90th percentile) as well as inter-individual coefficient of variation (COV, assessed by [SD/mean]) with approximately 15 participants in each age group: 18-30, 31-45, 46-60, and 60-70 years old. To assess intra-individual COV [assessed by [SD/mean]. To assess effect of standard diets containing 16.25 or 32.5 g fiber/day during the two 24 hour periods before and during the measurement of permeability
  Interventions: Other: Small Bowel and Colonic Permeability Test

INTERVENTIONS:
Other: Small Bowel and Colonic Permeability Test — small bowel and colonic permeability based on oral probe molecules and urine excretion in 60 healthy white, female and male adults aged 18-70y

SUMMARY:
To develop a test to measure small bowel and colonic permeability.

DETAILED DESCRIPTION:
The study consists of a physical examination, standardized meals and 3 oral sugar tests with 24 hour urine collections. It requires the participants to visit the Clinical Research Trials Unit in the Charlton Building and Domitilla Building. Remuneration will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-Obese
* Non-pregnant
* Caucasian
* BMI <30kg/m2

Exclusion Criteria:

* Diabetes
* Hypertension
* BMI ≥30kg/m2
* Chronic NSAID use (>3 days/week)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Standard Method to Measure Intestinal Permeability | 18 months
  Normal data on intestinal permeability in a Healthy human cohort:
  To summarize, using descriptive statistics, the median, 95% confidence interval, interquartile range of the following:
  * Urine excretion of probe molecules at 0-2h (reflecting small bowel permeability) with primary interest in 13C-mannitol and rhamnose
  * Urine excretion of probe molecules at 8-24h (reflecting colonic permeability) with primary interest in lactulose and sucralose
  * Urine excretion of probe molecules at 2-8h reflecting both small intestinal and colonic permeability As part of the effort to ascertain conditions under which the test would be performed in the future, we shall test the intra-individual coefficient of variation in healthy individuals, when the test is performed twice under conditions of identical diet, and when the test is performed with diets that have standardized but different quantities of fiber

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials